CLINICAL TRIAL: NCT02394912
Title: Evaluation of the Technical Success of Intravascular Ultrasound (IVUS) Guided Vena Cava Filter (VCF) Placement Using the LUMIFI™ With Crux® VCF System (LUMIFI Clinical Study)
Brief Title: Evaluation of the Technical Success of IVUS Guided VCF Placement Using the LUMIFI™ With Crux® VCF System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsatisfactory filter deployment in several cases
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140201
Record Dates: First submitted 2015-03-05; First posted 2015-03-20 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis
Keywords: vena cava filter
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

ARMS (1):
- Single-arm (Experimental)
  Interventions: Device: vena cava filter implantation (LUMIFI with Crux VCF System)

INTERVENTIONS:
Device: vena cava filter implantation (LUMIFI with Crux VCF System)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the LUMIFI with Crux VCF System for deployment of the Crux VCF. The study will compare the method of Crux VCF deployment using the LUMIFI with Crux VCF System (IVUS guidance) with the historical results of the Crux VCF System (fluoroscopic guidance). The study will include enrollment into a roll in phase consisting of 2 study subjects per site prior to enrollment into the primary treatment phase for primary analyses. The purpose of the roll in phase is to assure compliance with site training on the use of the investigational device and protocol workflow.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >18 years of age.
2. Patient or their legally authorized representative understands the research nature of the study and is willing and capable of providing informed consent
3. Patient has appropriate femoral vein access
4. Patient at risk for PE and meets at least one of the following sets of conditions:

   a. Documented DVT or PE and: i. Inability to anticoagulate the patient due to risk of bleeding such as recent surgery, trauma, intracranial bleed, GI bleed, OR ii. Progression/recurrence of DVT or PE on therapeutic anticoagulation, OR iii. Inability to anticoagulate due to high risk of tumor bleeding, OR iv. Patient unable to safely comply with anticoagulation, OR v. Patient that needs interruption of therapeutic anticoagulation such as at the time of an operation or other procedure.

   b. Patient that is high risk for DVT or PE and cannot be safely anticoagulated such as severe multi-trauma patient or patient having procedure with high risk for thromboembolism such as bariatric surgery.

   c. Patients with DVT at high risk for PE and free floating iliac or caval thrombosis d. Patients with compromised cardiopulmonary reserve from existing PE with right heart failure/strain who could not tolerate any further insult from new PE

Exclusion Criteria:

1. Patient has any one of the following conditions:

   1. Thrombus in the iliac veins or the IVC that precludes access to appropriate placement of the Crux Filter
   2. Known inadequate venous anatomy to allow insertion or retrieval of the filter from the IVC
   3. Known duplicated or left-sided IVC
   4. Known IVC transverse diameter at target lower renal ostia > 28mm or < 17mm
   5. Known extrinsic compression from abdominal or pelvic mass
   6. Known tumor thrombus involving the central venous system
   7. Uncontrolled sepsis, infection or persistent bacteremia
   8. Patient is at risk for septic pulmonary embolism
   9. Patient has an existing implanted filter in the IVC or superior vena cava (SVC) or underwent filter retrieval in previous 60 days.
   10. Patient has uncontrollable or active coagulopathy or known uncorrectable bleeding diathesis
   11. Patient has a condition that inhibits radiographic visualization of the IVC for post-deployment assessment
2. Patient has a known allergy or intolerance to polytetrafluoroethylene (PTFE) or Nitinol (nickel-titanium)
3. Patients unwilling or unable to comply with the protocol
4. Patients with history of or known reaction or sensitivity to contrast agent that cannot be pre-medicated
5. Female patient of childbearing potential who is pregnant (she must have negative pregnancy test within the 48 hours prior to implantation and any retrieval procedure)
6. Patient is participating in another device or drug clinical trial or has participated in such trial in the 30 days prior to enrollment
7. Investigator considers patient to be a poor candidate for the study or believes that the patient may compromise the study, e.g., concomitant conditions (reasons will be documented)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Jacobs, MD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - Surgical Care Associates, Louisville, Kentucky
  - Vascular Access Solutions, Orangeburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a prospective, single-arm, multicenter clinical study to evaluate the safety & effectiveness of the LUMIFI with Crux VCF system. The study included enrollment into a roll-in phase Cohort A consisting of 2 subjects/ site to assure compliance with the Investigational Device prior to enrolling into Cohort B, the treatment phase.
Groups:
- LUMIFI With Crux VCF System: vena cava filter implantation (LUMIFI with Crux VCF System). Includes both Cohort A and Cohort B subjects.
Period: Overall Study
Arm/Group | LUMIFI With Crux VCF System
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- LUMIFI With Crux VCF System: vena cava filter implantation (LUMIFI with Crux VCF System)
Arm/Group | LUMIFI With Crux VCF System
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Technical Success Rate
Description: All Subjects, Cohort A and Cohort B were included in the safety analysis. The primary endpoint of effectiveness, defined as technical success included only subjects within Cohort B. Technical success of filter placement is defined as the primary deployment of the filter such that the investigator judges the location to be suitable to provide sufficient mechanical protection against pulmonary embolism.
  Due to early stoppage of the study, enrollment of 100 subjects required to test the null hypothesis and evaluate the Primary Endpoint of Technical Success was not achieved. Therefore, a formal analysis of Technical Success was not performed.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Roll-in phase consisting of 2 subjects per site to assure compliance with use of the Investigational Device
- Cohort B: Subjects are enrolled into Cohort B after each site has enrolled 2 subjects in Cohort A to assure compliance with use of the Investigational Device
Arm/Group | LUMIFI With Crux VCF System | Cohort A | Cohort B
Number analyzed (Participants) | 21 | 8 | 13
Participants | 16 | 6 | 10

ADVERSE EVENTS:
Arm/Group | LUMIFI With Crux VCF System
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUMIFI With Crux VCF System (N=21)
Pulmonary Emboli Bilaterial (Vascular disorders) | 1 (1)
Filter deployed too low (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator shall have the right to publish or otherwise make public any data resulting from the study upon the earlier of (a) publication of a multi-center publication (or any publication, if the Study is not a multi-center study) coordinated by Sponsor with respect to the data resulting from the study, and (b) eighteen (18) months after the Study is completed at all participating sites if a multi-center publication.